CLINICAL TRIAL: NCT05896761
Title: Sub-study to the A2M Study to Evaluate the Pharmacokinetics, Tolerability and Efficacy of Cabotegravir and Rilpivirine Long-Acting Injections Following Intramuscular Administration in the Vastus Lateralis Muscle (Thigh) in HIV-infected Adult Participants Who Have Received at Least Three Years of Gluteal Injections in the A2M Study
Brief Title: A Sub-study of Cabotegravir (CAB) and Rilpivirine (RPV) in Human Immunodeficiency Viruses (HIV)-Infected Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207966-001
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Human Immunodeficiency Virus Type 1 (HIV-1)
Keywords: Cabotegravir; Efficacy; Human immunodeficiency virus; Pharmacokinetic; Rilpivirine; Safety; Tolerability
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving CAB LA 400 milligrams (mg) and RPV LA 600 mg (Experimental): Participants will receive an Intramuscular (IM) injection of CAB LA 400 mg on one lateral thigh and RPV LA 600 mg into the opposite lateral thigh on Day 1 in every 4 weeks (Q4W) for a total of 16 weeks during Thigh injection phase. Participants will then return to the clinic 4 weeks later to receive their first IM gluteal injection (at Week 16) of CAB LA 400 mg and RPV LA 600 mg during the Return to Gluteal Injection Phase. The subsequent gluteal injection will occur at Week 20.
  Interventions: Drug: Cabotegravir Injectable Suspension; Drug: Rilpivirine Injectable Suspension
- Participants receiving CAB LA 600 mg and RPV LA 900 mg (Experimental): Participants will receive an IM injection of CAB LA 600 mg on one lateral thigh and RPV LA 900 mg into the opposite lateral thigh on Day 1 in every 8 weeks (Q8W) for a total of 16 weeks during Thigh injection phase. Participants will then return to the clinic 8 weeks later receive their first IM gluteal injection (at Week 16) of CAB LA 600mg and RPV LA 900 mg during the Return to Gluteal Injection phase. The subsequent gluteal injection will occur at Week 24.
  Interventions: Drug: Cabotegravir Injectable Suspension; Drug: Rilpivirine Injectable Suspension

INTERVENTIONS:
Drug: Cabotegravir Injectable Suspension — CAB LA injectable suspension is a sterile white to slightly pink suspension containing 200 milligrams per milliliter (mg/mL) of GSK1265744 as free acid for administration by IM injection. CAB LA injectable suspension is to be stored at up to 30 degree Celsius and should not be frozen.
Drug: Rilpivirine Injectable Suspension — RPV LA injectable suspension is a sterile white suspension containing 300 mg/mL of RPV as the free base for administration by IM injection. RPV LA injectable suspension should be kept in the outer package and stored at 2-8 degree Celsius and should not be frozen. RPV LA should also be protected from light.

SUMMARY:
This sub-study will assess the pharmacokinetics (PK), safety, tolerability, virologic efficacy and health outcomes of CAB (GSK1265744) and RPV long acting (LA) in HIV-infected adult participants currently enrolled in the Antiretroviral Therapy as Long Acting Suppression every 2 Months (ATLAS2M [A2M]) study (NCT03299049).

ELIGIBILITY:
Inclusion Criteria:

Sub-study specific Inclusion Criteria:

* Capable of giving sub-study specific informed consent.
* Eligible participants must have been on CAB LA + RPV LA regimen for a minimum of 152 weeks while on the ATLAS2-M study. Any disruptions in dosing during ATLAS2-M must be discussed with the Medical Monitor for a final determination of eligibility into the sub-study.
* Plasma HIV-1 RNA <50 copies/mL at Sub-Study Screening.

Inclusion criteria detailed for the ATLAS-2M main study apply to the sub-study:

* A female participant is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotropin [hCG] test) not lactating, and at least one of the following conditions applies:

  1. Non-reproductive potential defined as:

     * Pre-menopausal females with one of the following:

       i. Documented tubal ligation ii. Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion iii. Hysterectomy iv. Documented Bilateral Oophorectomy
     * Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.
  2. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, throughout the study, for at least 30 days after discontinuation of all oral study medications, and for at least 52 weeks after discontinuation of CAB LA and RPV LA.
* The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception.

Exclusion Criteria:

Sub-study specific Exclusion Criteria:

* Participants with more than 1 plasma HIV-1 RNA measurement >=50 copies/mL to <200 copies/mL (virologic blip) within 24 weeks prior to sub-study Screening visit.
* Any Suspected Virologic Failure (HIV-RNA greater than [>]200 copies/mL as defined in during ATLAS-2M study.
* Participants planning to require oral bridging during participation in the ATLAS-2M sub-study.
* The participant has a tattoo or any dermatological condition overlying the thigh region which may interfere with interpretation of injection site reactions.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.

Exclusion criteria detailed for the ATLAS-2M main study apply to the sub-study:

* Women who are pregnant, breastfeeding or plan to become pregnant or breastfeed during the study.
* Any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy, and Cluster of Differentiation 4 positive (CD4+) counts <200 cells per microliter are not exclusionary.
* Participants with moderate to severe hepatic impairment.
* Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrollment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrollment.
* Participants who, in the investigator's judgment, pose a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis.
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the participant prior to randomization.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during PK sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled.
* Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid lesser than or equal to (<=)325 mg or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease.
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening phase to verify a result.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound.
* Participant has estimated creatine clearance <50mL per minute per 1.73 square meter via Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) Method.
* Alanine aminotransferase (ALT) >=3 × upper limit of normal (ULN) at Screening.
* Exposure to an experimental drug (with the exception of those in the ATLAS-2M study including CAB, CAB LA, and RPV, RPV LA) or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study.
* Treatment with any of the following agents within 28 days of Screening:

  i. radiation therapy; ii. cytotoxic chemotherapeutic agents; iii. tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid [INH]); iv. anti-coagulation agents; v. Immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Use of medications which are associated with Torsade de Pointes.
* Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (30):
- United States (10):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Lynchburg, Virginia
- Argentina (2):
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
- Canada (2):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Regina, Saskatchewan
- Germany (4):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Milan, Lombardy, Italy
- Spain (9):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a sub-study of Cabotegravir (CAB) and Rilpivirine (RPV) long-acting (LA) in Human Immunodeficiency Viruses (HIV)-infected participants currently enrolled in the Antiretroviral Therapy as Long- Acting Suppression every 2 Months (ATLAS2M [A2M]) study (NCT03299049).
Pre-assignment Details: A total of 118 participants were enrolled in the study.
Groups:
- CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W): Participants received an intramuscular (IM) injection of CAB LA 600 mg on one lateral thigh and RPV LA 900 mg into the opposite lateral thigh on Day 1 in every 8 weeks (Q8W) for a total of 16 weeks during Thigh Injection Phase. Participants then returned to the clinic 8 weeks later to receive first IM gluteal injection (at Week 16) of CAB LA 600 mg + RPV LA 900 mg during the Return to Gluteal (Glu) Injection (Inj) Phase and subsequent gluteal injection occurred after Q8W.
- CAB LA 400 mg + RPV LA 600 mg (Q4W): Participants received an IM injection of CAB LA 400 mg on one lateral thigh and RPV LA 600 mg into the opposite lateral thigh on Day 1 in every 4 weeks (Q4W) for a total of 16 weeks during Thigh Injection Phase. Participants then returned to the clinic 4 weeks later received first IM gluteal injection (at Week 16) of CAB LA 400 mg + RPV LA 600 mg during the Return to Gluteal Injection Phase and subsequent gluteal injection occurred after Q4W.
Period: Thigh Injection Phase (Up to Week 16)
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Started | 54 | 64
Completed | 51 | 61
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Period: Return to Glu Inj Phase (Weeks 16 to 24)
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Started | 51 | 61
Completed | 51 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W) | Total
Number analyzed (Participants) | 54 | 64 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (12.56) | 46.6 (10.60) | 47.5 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 26 | 45
  Male | 35 | 38 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 1 | 1
  ASIAN - JAPANESE HERITAGE | 0 | 1 | 1
  BLACK OR AFRICAN AMERICAN | 11 | 7 | 18
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 43 | 54 | 97
  MULTIPLE | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Concentration at End of Dosing Interval (Ctau) of CAB LA Following Administration of CAB LA + RPV LA Q8W
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis.
Time Frame: Weeks -8,-7,-4 and Pre-dose on Day 1(Pre-Thigh Gluteal Injection);2 Hours post-dose on Day 1,Pre-dose on Week 8,Weeks 1 and 4 post-dose(First Thigh Injection);2 Hours post-dose on Week 8 and Weeks 9, 12 post-dose,Pre-dose on Week 16(Last Thigh Injection)
Population: Sub-study pharmacokinetic (PK) parameter Population included all participants who received at least one CAB and/or RPV thigh injection and had at least one evaluable PK parameter estimate during the sub-study. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- CAB+RPV Q8W First Thigh Injection: Participants received a first IM injection of CAB LA 600 mg on one lateral thigh and RPV LA 900 mg into the opposite lateral thigh on Day 1 during Thigh Injection Phase.
- CAB+RPV Q8W Last Thigh Injection: Participants received an IM injection of CAB LA 600 mg on one lateral thigh and RPV LA 900 mg into the opposite lateral thigh on Week 8 during Thigh Injection Phase.
- CAB+RPV Q8W Pre-Thigh Gluteal Injection: Participants received an IM gluteal injections of CAB LA 600 mg and RPV LA 900 mg at Week -8 during Pre-Thigh Gluteal Injection Phase.
Arm/Group | CAB+RPV Q8W First Thigh Injection | CAB+RPV Q8W Last Thigh Injection | CAB+RPV Q8W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 40 | 36 | 40
Micrograms per milliliter | 1.67 (69.3) | 1.61 (55.5) | 1.81 (51.6)
Statistical Analysis 1: Comparison: CAB+RPV Q8W First Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 0.926, 90% CI 2-sided [0.831 to 1.03]
Statistical Analysis 2: Comparison: CAB+RPV Q8W Last Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 0.929, 90% CI 2-sided [0.816 to 1.06]

2. Primary Outcome: Concentration at End of Dosing Interval (Ctau) of RPV LA Following Administration of CAB LA + RPV LA Q8W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 1
Population: Sub-study PK parameter Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | CAB+RPV Q8W First Thigh Injection | CAB+RPV Q8W Last Thigh Injection | CAB+RPV Q8W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 40 | 36 | 40
Nanograms per milliliter | 103 (49.7) | 117 (54.1) | 104 (41.5)
Statistical Analysis 1: Comparison: CAB+RPV Q8W First Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.06, 90% CI 2-sided [0.966 to 1.17]
Statistical Analysis 2: Comparison: CAB+RPV Q8W Last Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.18, 90% CI 2-sided [1.07 to 1.29]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of CAB LA Following Administration of CAB LA + RPV LA Q8W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB+RPV Q8W First Thigh Injection | CAB+RPV Q8W Last Thigh Injection | CAB+RPV Q8W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 54 | 50 | 54
Micrograms per milliliter | 4.52 (37.7) | 3.70 (40.8) | 3.36 (41.4)
Statistical Analysis 1: Comparison: CAB+RPV Q8W First Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.35, 90% CI 2-sided [1.22 to 1.49]
Statistical Analysis 2: Comparison: CAB+RPV Q8W Last Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.10, 90% CI 2-sided [0.975 to 1.24]

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of RPV LA Following Administration of CAB LA + RPV LA Q8W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | CAB+RPV Q8W First Thigh Injection | CAB+RPV Q8W Last Thigh Injection | CAB+RPV Q8W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 54 | 51 | 54
Nanograms per milliliter | 184 (33.9) | 172 (47.4) | 146 (56.5)
Statistical Analysis 1: Comparison: CAB+RPV Q8W First Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.26, 90% CI 2-sided [1.12 to 1.40]
Statistical Analysis 2: Comparison: CAB+RPV Q8W Last Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.18, 90% CI 2-sided [1.09 to 1.28]

5. Primary Outcome: Area Under the Concentration Curve From 0 Hours to the Time of Next Dosing (AUC [0-tau]) of CAB LA Following Administration of CAB LA + RPV LA Q8W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram/milliliter
Arm/Group | CAB+RPV Q8W First Thigh Injection | CAB+RPV Q8W Last Thigh Injection | CAB+RPV Q8W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 48 | 38 | 47
Hour*microgram/milliliter | 4038 (34.6) | 3384 (36.6) | 3344 (32.9)
Statistical Analysis 1: Comparison: CAB+RPV Q8W First Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.21, 90% CI 2-sided [1.13 to 1.30]
Statistical Analysis 2: Comparison: CAB+RPV Q8W Last Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.09, 90% CI 2-sided [1.00 to 1.20]

6. Primary Outcome: Area Under the Concentration Curve From 0 Hours to the Time of Next Dosing (AUC [0-tau]) of RPV LA Following Administration of CAB LA + RPV LA Q8W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter
Arm/Group | CAB+RPV Q8W First Thigh Injection | CAB+RPV Q8W Last Thigh Injection | CAB+RPV Q8W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 48 | 39 | 47
Hour*nanogram/milliliter | 179483 (33.8) | 190641 (50.4) | 162046 (36.7)
Statistical Analysis 1: Comparison: CAB+RPV Q8W First Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.15, 90% CI 2-sided [1.07 to 1.23]
Statistical Analysis 2: Comparison: CAB+RPV Q8W Last Thigh Injection vs CAB+RPV Q8W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.29, 90% CI 2-sided [1.20 to 1.38]

7. Primary Outcome: Concentration at End of Dosing Interval (Ctau) of CAB LA Following Administration of CAB LA + RPV LA Q4W
Description: Blood samples were collected for PK analysis.
Time Frame: Weeks -4 and -3, Pre-dose on Day 1 (Pre-Thigh Gluteal Injection); 2 Hours post-dose on Day 1, Week 1 post-dose, Pre-dose on Week 4 (First Thigh Injection); 2 Hours post-dose on Week 12, Week 13 post-dose and Pre-dose on Week 16 (Last Thigh Injection)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- CAB+RPV Q4W First Thigh Injection: Participants received a first IM injection of CAB LA 400 mg on one lateral thigh and RPV LA 600 mg into the opposite lateral thigh on Day 1 during Thigh Injection Phase.
- CAB+RPV Q4W Last Thigh Injection: Participants received an IM injection of CAB LA 400 mg on one lateral thigh and RPV LA 600 mg into the opposite lateral thigh on Week 12 during Thigh Injection Phase.
- CAB+RPV Q4W Pre-Thigh Gluteal Injection: Participants received an IM gluteal injections of CAB LA 400 mg and RPV LA 600 mg at Week -4 during Pre-Thigh Gluteal Injection Phase.
Arm/Group | CAB+RPV Q4W First Thigh Injection | CAB+RPV Q4W Last Thigh Injection | CAB+RPV Q4W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 53 | 52 | 52
Micrograms per milliliter | 3.34 (34.6) | 3.00 (37.8) | 2.94 (38.9)
Statistical Analysis 1: Comparison: CAB+RPV Q4W First Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.16, 90% CI 2-sided [1.08 to 1.25]
Statistical Analysis 2: Comparison: CAB+RPV Q4W Last Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 0.983, 90% CI 2-sided [0.890 to 1.09]

8. Primary Outcome: Concentration at End of Dosing Interval (Ctau) of RPV LA Following Administration of CAB LA + RPV LA Q4W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | CAB+RPV Q4W First Thigh Injection | CAB+RPV Q4W Last Thigh Injection | CAB+RPV Q4W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 53 | 52 | 52
Nanograms per milliliter | 170 (35.2) | 171 (39.8) | 162 (37.6)
Statistical Analysis 1: Comparison: CAB+RPV Q4W First Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.06, 90% CI 2-sided [0.991 to 1.13]
Statistical Analysis 2: Comparison: CAB+RPV Q4W Last Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.04, 90% CI 2-sided [0.974 to 1.12]

9. Primary Outcome: Maximum Plasma Concentration (Cmax) of CAB LA Following Administration of CAB LA + RPV LA Q4W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB+RPV Q4W First Thigh Injection | CAB+RPV Q4W Last Thigh Injection | CAB+RPV Q4W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 61 | 59 | 63
Micrograms per milliliter | 4.65 (38.3) | 4.09 (35.6) | 3.95 (35.8)
Statistical Analysis 1: Comparison: CAB+RPV Q4W First Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.18, 90% CI 2-sided [1.11 to 1.25]
Statistical Analysis 2: Comparison: CAB+RPV Q4W Last Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.06, 90% CI 2-sided [0.989 to 1.14]

10. Primary Outcome: Maximum Plasma Concentration (Cmax) of RPV LA Following Administration of CAB LA + RPV LA Q4W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | CAB+RPV Q4W First Thigh Injection | CAB+RPV Q4W Last Thigh Injection | CAB+RPV Q4W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 62 | 59 | 63
Nanograms per milliliter | 210 (34.9) | 205 (34.8) | 197 (33.8)
Statistical Analysis 1: Comparison: CAB+RPV Q4W First Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.08, 90% CI 2-sided [1.03 to 1.12]
Statistical Analysis 2: Comparison: CAB+RPV Q4W Last Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.04, 90% CI 2-sided [0.997 to 1.08]

11. Primary Outcome: Area Under the Concentration Curve From 0 Hours to the Time of Next Dosing (AUC [0-tau]) of CAB LA Following Administration of CAB LA + RPV LA Q4W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | CAB+RPV Q4W First Thigh Injection | CAB+RPV Q4W Last Thigh Injection | CAB+RPV Q4W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 54 | 55 | 58
Hours*micrograms per milliliter | 2558 (34.4) | 2379 (34.8) | 2275 (35.1)
Statistical Analysis 1: Comparison: CAB+RPV Q4W First Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.13, 90% CI 2-sided [1.08 to 1.19]
Statistical Analysis 2: Comparison: CAB+RPV Q4W Last Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.04, 90% CI 2-sided [0.97 to 1.11]

12. Primary Outcome: Area Under the Concentration Curve From 0 Hours to the Time of Next Dosing (AUC [0-tau]) of RPV LA Following Administration of CAB LA + RPV LA Q4W
Description: Blood samples were collected for PK analysis.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | CAB+RPV Q4W First Thigh Injection | CAB+RPV Q4W Last Thigh Injection | CAB+RPV Q4W Pre-Thigh Gluteal Injection
Number analyzed (Participants) | 55 | 55 | 58
Hour*nanogram per milliliter | 120963 (32.6) | 123197 (33.6) | 115202 (33.9)
Statistical Analysis 1: Comparison: CAB+RPV Q4W First Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.06, 90% CI 2-sided [1.02 to 1.11]
Statistical Analysis 2: Comparison: CAB+RPV Q4W Last Thigh Injection vs CAB+RPV Q4W Pre-Thigh Gluteal Injection; Test type: Other; Ratio of geometric least square mean = 1.06, 90% CI 2-sided [1.01 to 1.11]

13. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs) by Maximum Severity Grade - Thigh Injection Phase
Description: Severity of ISRs was analyzed using division of acquired immunodeficiency syndrome (DAIDS) grading scale. The severity is categorized into grades as following: Grade 1 - mild, Grade 2 - moderate, Grade 3 - severe, Grade 4 - Potentially life threatening, Grade 5 - Death. Higher grade indicates more severe condition. Data for number of participants with maximum grade or intensity for overall ISRs were reported.
Time Frame: Up to Week 16
Population: Sub-study Safety Population included all randomized participants who received at least one CAB and/or RPV thigh injection. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 38 | 45
Participants
  Mild or Grade 1 | 18 | 27
  Moderate or Grade 2 | 16 | 12
  Severe or Grade 3 | 4 | 6
  Potentially Life-Threatening or Grade 4 | 0 | 0
  Death or Grade 5 | 0 | 0

14. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) Based on Maximum Severity Grade- Thigh Injection Phase
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Severity of AESI was analyzed using DAIDS grading scale. The severity is categorized into grades as following: Grade 1 - mild, Grade 2 - moderate, Grade 3 - severe, Grade 4 - Potentially life threatening, Grade 5 - Death. Higher grade indicates more severe condition. Data for number of participants with common AESI based on maximum severity were reported.
Time Frame: Up to Week 16
Population: Sub-study Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 38 | 45
Participants
  Mild or Grade 1 | 18 | 27
  Moderate or Grade 2 | 16 | 12
  Severe or Grade 3 | 4 | 6
  Potentially Life-Threatening or Grade 4 | 0 | 0
  Death or Grade 5 | 0 | 0

15. Secondary Outcome: Number of Participants Who Discontinue Treatment Due to ISRs and AESIs-Thigh Injection Phase
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants who discontinued treatment due to ISRs and AESIs is presented.
Time Frame: Up to Week 16
Population: Sub-study Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 54 | 64
Participants
  Discontinuations due to AESI | 1 | 0
  Discontinuations due to ISR | 1 | 0

16. Secondary Outcome: Percentage of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) Less Than (<)50 Copies Per Milliliter (Copies/mL) Using the Food and Drug (FDA) Snapshot Algorithm-Thigh Injection Phase
Description: Percentage of participants with plasma HIV-1 RNA < 50 copies/mL was obtained using the FDA snapshot algorithm. Baseline was the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Percentage values are rounded off.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16
Population: Sub-study Intent-to-treat Exposed Population included all randomized participants who received at least one CAB and/or RPV thigh injection.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 54 | 64
Percentage of participants
  Baseline (Day 1) | 100 [93 to 100] | 98 [95 to 100]
  Week 4 | 100 [93 to 100] | 98 [95 to 100]
  Week 8 | 96 [91 to 100] | 97 [93 to 100]
  Week 12 | 94 [88 to 100] | 95 [90 to 100]
  Week 16 | 94 [88 to 100] | 95 [90 to 100]

17. Secondary Outcome: Percentage of Participants With Plasma HIV RNA Greater Than or Equal to (>=)50 Copies/mL Over Time as Per the FDA Snapshot Algorithm- Thigh Injection Phase
Description: Percentage of participants with plasma HIV 1 RNA >= 50 copies/mL was obtained using the FDA snapshot algorithm. Baseline was the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Percentage values are rounded off.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16
Population: Sub-study Intent-to-Treat Exposed Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 54 | 64
Percentage of participants
  Baseline (Day 1) | 0 [0.0 to 6.6] | 1.6 [0.0 to 4.6]
  Week 4 | 0 [0.0 to 6.6] | 0 [0.0 to 5.6]
  Week 8 | 0 [0.0 to 6.6] | 0 [0.0 to 5.6]
  Week 12 | 0 [0.0 to 6.6] | 0 [0.0 to 5.6]
  Week 16 | 0 [0.0 to 6.6] | 0 [0.0 to 5.6]

18. Secondary Outcome: Percentage of Participants With Protocol-defined Confirmed Virologic Failure (CVF)- Thigh Injection Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. CVF was defined as rebound as indicated by two consecutive plasma HIV-1-RNA levels >=200 copies/mL after prior suppression to <200 copies/mL. Percentage of participants with protocol-defined CVF were reported.
Time Frame: Up to Week 16
Population: Sub-study Intent-to-treat Exposed Population
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 54 | 64
Percentage of participants | 0 | 0

19. Secondary Outcome: Number of Participants With Treatment Emergent Genotypic Resistance - Thigh Injection Phase
Description: Plasma samples were collected for drug resistance testing. Number of participants who met CVF criteria (two consecutive plasma HIV-1-RNA levels >=200 copies/mL after prior suppression to <200 copies/mL) with treatment emergent genotypic resistance were reported.
Time Frame: Up to Week 16
Population: Sub-study Confirmed Virologic Failure Population comprised of all participants who received at least one CAB and/or RPV thigh injection who met Confirmed Virologic Failure (CVF) criteria in the sub-study. Only participants with CVF were included in the analysis.
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Participants With Treatment Emergent Phenotypic Resistance - Thigh Injection Phase
Description: Plasma samples were collected for drug resistance testing. Number of participants who met CVF criteria (two consecutive plasma HIV-1-RNA levels >=200 copies/mL after prior suppression to <200 copies/mL) with treatment emergent phenotypic resistance were reported.
Time Frame: Up to Week 16
Population: Sub-study Confirmed Virologic Failure Population. Only participants with CVF were included in the analysis.
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Number of Participants With Post-injection Pain Using Numerical Rating Scale (NRS) on Day 1-Thigh Injection Phase
Description: A numeric rating scale was used to assess the level of pain experienced following injections with CAB + RPV. The scale contains one item and the response scale is ranging from 0= "no pain" to 10= "extreme pain". NRS questionnaire included two questions regarding the maximum level of pain experienced with the most recent injections.
Time Frame: Day 1
Population: Sub-study Intent-to-Treat Exposed Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 54 | 64
Participants
  Score 0 | 14 | 21
  Score 1 | 13 | 16
  Score 2 | 7 | 6
  Score 3 | 6 | 7
  Score 4 | 5 | 4
  Score 5 | 4 | 4
  Score 6 | 3 | 2
  Score 7 | 0 | 3
  Score 8 | 1 | 0
  Score 9 | 1 | 0
  Score 10 | 0 | 1

22. Secondary Outcome: Number of Participants With Post-injection Pain Using Numerical Rating Scale (NRS) for CAB LA + RPV LA Q8W Arm on Week 8- Thigh Injection Phase
Description: as for outcome 21
Time Frame: Week 8
Population: Sub-study Intent-to-Treat Exposed Population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W): Participants received an intramuscular (IM) injection of CAB LA 600 mg on one lateral thigh and RPV LA 900 mg into the opposite lateral thigh on Day 1 in every 8 weeks (Q8W) for a total of 16 weeks during thigh injection phase. Participants then returned to the clinic 8 weeks later to receive first IM gluteal injection (at Week 16) of CAB LA 600 mg + RPV LA 900 mg during the return to gluteal injection phase and subsequent gluteal injection occurred after Q8W.
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W)
Number analyzed (Participants) | 51
Participants
  Score 0 | 15
  Score 1 | 11
  Score 2 | 9
  Score 3 | 5
  Score 4 | 1
  Score 5 | 3
  Score 6 | 2
  Score 7 | 2
  Score 8 | 1
  Score 9 | 1
  Score 10 | 1

23. Secondary Outcome: Number of Participants With Post-injection Pain Using Numerical Rating Scale (NRS) for CAB LA + RPV LA Q4W Arm on Week 12- Thigh Injection Phase
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 61
Participants
  Score 0 | 20
  Score 1 | 12
  Score 2 | 7
  Score 3 | 4
  Score 4 | 9
  Score 5 | 4
  Score 6 | 1
  Score 7 | 1
  Score 8 | 0
  Score 9 | 2
  Score 10 | 1

24. Secondary Outcome: Number of Participants With Post-injection Pain Using Numerical Rating Scale (NRS)- Return to Gluteal Injection Phase
Description: as for outcome 21
Time Frame: Study Week 16
Population: Sub-study Intent-to-Treat Exposed Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 51 | 61
Participants
  Score 0 | 14 | 22
  Score 1 | 8 | 11
  Score 2 | 10 | 6
  Score 3 | 6 | 8
  Score 4 | 5 | 3
  Score 5 | 1 | 2
  Score 6 | 5 | 5
  Score 7 | 1 | 0
  Score 8 | 0 | 3
  Score 9 | 1 | 1
  Score 10 | 0 | 0

25. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Status Version (HIVTSQs) Total Score at Indicated Time Points-Thigh Injection Phase
Description: HIVTSQ is a self-completion measure specifically designed to measure treatment satisfaction in HIV participants. HIVTSQs questionnaire comprises 1-12 questions and the total treatment satisfaction score is computed with items 1-11 and summed to produce a total score with a possible range of 0 to 66. Higher scores indicate a greater satisfaction and a lower score indicate dissatisfaction. Baseline was the latest pre-treatment assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 54 | 64
Scores on a scale
  Baseline (Day 1) | 63.85 (3.378) | 64.03 (3.376)
  Week 16: number analyzed (Participants) | 51 | 61
  Week 16 | 61.69 (6.912) | 61.74 (8.786)

26. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Status Version (HIVTSQs) Total Score at Indicated Time Points for CAB LA + RPV LA Q8W Arm -Return to Gluteal Injection Phase
Description: HIVTSQ is a self-completion measure specifically designed to measure treatment satisfaction in HIV participants. HIVTSQs questionnaire comprises 1-12 questions and the total treatment satisfaction score is computed with items 1-11 and summed to produce a score with a possible range of 0 to 66. Higher scores indicate a greater satisfaction and a lower score indicate dissatisfaction.
Time Frame: Study Week 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W)
Number analyzed (Participants) | 51
Scores on a scale | 63.78 (3.743)

27. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Status Version (HIVTSQs) Total Score at Indicated Time Points for CAB LA + RPV LA Q4W Arm -Return to Gluteal Injection Phase
Description: as for outcome 26
Time Frame: Study Week 20
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 61
Scores on a scale | 63.25 (4.911)

28. Secondary Outcome: Change From Baseline in HIV Treatment Satisfaction Questionnaire - Status Version (HIVTSQs) Individual Item Score at Indicated Time Points- Thigh Injection Phase
Description: HIVTSQs is a 12-item questionnaire and individual item scores on HIVTSQs scale are rated as 6(very satisfied) to 0(very dissatisfied).Higher scores represent greater satisfaction.Data was reported for each treatment satisfaction item based on(Item1=satisfaction with current treatment,Item2=level of HIV control based on treatment,Item3=any side effects of present treatment,Item4=demands made by current treatment,Item5=convenience in finding treatment,Item6=flexibility in finding treatment,Item7=understanding HIV,Item8=extent to which the treatment fits in with lifestyle, Item9=recommendation of present treatment to someone else,Item10=continuation with present form of treatment,Item11=easy or difficult treatment,Item12=amount of discomfort/pain involved with present form of treatment).Baseline was latest pre-treatment assessment with a non-missing value, including those from unscheduled visits.Change from Baseline was calculated by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline (Day 1) and up to Week 16
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 51 | 61
Scores on a scale
  Item 1 | -0.3 (1.37) | -0.3 (1.09)
  Item 2 | -0.1 (0.27) | 0.0 (0.38)
  Item 3 | -0.7 (1.32) | -0.2 (0.92)
  Item 4 | -0.2 (0.81) | -0.2 (0.96)
  Item 5 | -0.1 (0.63) | -0.2 (0.87)
  Item 6 | 0.0 (0.88) | -0.3 (0.86)
  Item 7 | -0.1 (0.73) | -0.1 (0.64)
  Item 8 | -0.1 (0.95) | -0.1 (0.84)
  Item 9 | -0.2 (0.92) | -0.1 (0.83)
  Item 10 | -0.3 (1.11) | -0.3 (1.12)
  Item 11 | -0.1 (0.83) | -0.4 (1.02)
  Item 12 | -0.7 (1.87) | -0.5 (1.29)

29. Secondary Outcome: Change From Study Week 16 to Study Week 24 in HIV Treatment Satisfaction Questionnaire - Status Version (HIVTSQs) Individual Item Score at Indicated Time Points for CAB LA + RPV LA Q8W Arm- Return to Gluteal Injection
Description: HIVTSQs is a 12-item questionnaire and individual item scores on HIVTSQs scale are rated as 6 (very satisfied) to 0 (very dissatisfied). Higher scores represent greater satisfaction with each aspect of treatment. Data was reported for each treatment satisfaction item based on (Item 1=satisfaction with current treatment, Item 2=level of HIV control based on treatment, Item 3=any side effects of present treatment, Item 4=demands made by current treatment, Item 5=convenience in finding treatment, Item 6=flexibility in finding treatment, Item 7=understanding HIV, Item 8=extent to which the treatment fits in with lifestyle, Item 9=recommendation of present treatment to someone else, Item 10=continuation with present form of treatment, Item 11=easy or difficult treatment, Item 12=amount of discomfort/pain involved with present form of treatment). Change from Study Week 16 to Study Week 24 was calculated by subtracting the Study Week 16 value from the Study Week 24 value.
Time Frame: Study Week 16 and Study Week 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W)
Number analyzed (Participants) | 51
Scores on a scale
  Item 1 | 0.3 (1.16)
  Item 2 | 0.0 (0.34)
  Item 3 | 0.5 (1.19)
  Item 4 | 0.2 (0.80)
  Item 5 | 0.1 (0.59)
  Item 6 | 0.3 (0.56)
  Item 7 | 0.0 (0.40)
  Item 8 | 0.2 (0.86)
  Item 9 | 0.2 (0.88)
  Item 10 | 0.2 (1.14)
  Item 11 | 0.1 (0.84)
  Item 12 | 0.7 (1.47)

30. Secondary Outcome: Change From Study Week 16 to Study Week 20 in HIV Treatment Satisfaction Questionnaire - Status Version (HIVTSQs) Individual Item Score at Indicated Time Points for CAB LA + RPV LA Q4W Arm- Return to Gluteal Injection Phase
Description: HIVTSQs is a 12-item questionnaire and individual item scores on HIVTSQs scale are rated as 6(very satisfied) to 0(very dissatisfied).Higher scores represent greater satisfaction.Data was reported for each treatment satisfaction item based on(Item1=satisfaction with current treatment,Item2=level of HIV control based on treatment,Item3=any side effects of present treatment,Item4=demands made by current treatment,Item5=convenience in finding treatment,Item6=flexibility in finding treatment,Item7=understanding HIV,Item8=extent to which the treatment fits in with lifestyle, Item9=recommendation of present treatment to someone else,Item10=continuation with present form of treatment,Item11=easy or difficult treatment,Item12=amount of discomfort/pain involved with present form of treatment).Change from Study Week 16 to Study Week 20 was calculated by subtracting the Study Week 16 value from the Study Week 20 value.
Time Frame: Study Week 16 and Study Week 20
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 61
Scores on a scale
  Item 1 | 0.2 (0.73)
  Item 2 | 0.1 (0.31)
  Item 3 | 0.3 (0.85)
  Item 4 | 0.1 (0.60)
  Item 5 | 0.1 (0.69)
  Item 6 | 0.1 (0.73)
  Item 7 | 0.0 (0.64)
  Item 8 | 0.0 (0.52)
  Item 9 | 0.1 (0.69)
  Item 10 | 0.2 (0.80)
  Item 11 | 0.3 (0.79)
  Item 12 | 0.4 (1.02)

31. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Change Version (HIVTSQc) Total Score at Indicated Time Points- Thigh Injection Phase
Description: HIVTSQ is a self-completion measure specifically designed to measure treatment satisfaction in HIV participants. Total treatment satisfaction change score is computed using items 1 to 11 and are summed to produce a score with a possible range of -33 to 33. Higher the score, greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of 0 represented no change.
Time Frame: Up to Week 16
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 51 | 61
Scores on a scale | 17.8 (16.02) | 19.7 (15.45)

32. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Change Version (HIVTSQc) Individual Item Score at Indicated Time Points- Thigh Injection Phase
Description: HIVTSQc is a 12-item questionnaire to measure treatment satisfaction in HIV participants. Individual items were rated as +3 (much more satisfied) to -3 (much less satisfied). Higher the score, greater the improvement in satisfaction with each aspect of treatment and lower the score, greater the deterioration in satisfaction with each aspect of treatment. Data was reported for each treatment satisfaction item based on (Item 1=satisfaction with current treatment, Item 2=level of HIV control based on treatment, Item 3=any side effects of present treatment, Item 4=demands made by current treatment, Item 5=convenience in finding treatment, Item 6=flexibility in finding treatment, Item 7=understanding HIV, Item 8=extent to which the treatment fits in with lifestyle, Item 9=recommendation of present treatment to someone else, Item 10=continuation with present form of treatment, Item 11=easy or difficult treatment, Item 12=amount of discomfort/pain involved with present form of treatment).
Time Frame: Up to Week 16
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W) | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 51 | 61
Scores on a scale
  Item 1 | 1.5 (1.84) | 1.7 (1.71)
  Item 2 | 1.8 (1.42) | 1.9 (1.42)
  Item 3 | 1.3 (1.92) | 1.5 (1.70)
  Item 4 | 1.5 (1.74) | 1.8 (1.48)
  Item 5 | 1.7 (1.53) | 1.6 (1.66)
  Item 6 | 1.6 (1.37) | 1.7 (1.50)
  Item 7 | 1.7 (1.44) | 2.0 (1.35)
  Item 8 | 1.7 (1.55) | 2.0 (1.47)
  Item 9 | 1.7 (1.80) | 2.0 (1.57)
  Item 10 | 1.5 (2.00) | 1.9 (1.71)
  Item 11 | 1.6 (1.69) | 1.7 (1.65)
  Item 12 | 1.0 (2.14) | 1.4 (1.74)

33. Secondary Outcome: Number of Participants With Their Treatment Preference as Assessed Using Preference Questionnaire for CAB LA + RPV LA Q8W Arm
Description: A preference questionnaire was used to assess participant's preference for the thigh injections compared with the gluteal injections. The "Preference" questionnaire included a single item question evaluating preference of HIV treatment. Participants were required to provide their response to Question, which stated "Which injection site do you prefer". The responses included Injections in the buttock, Injections in the thigh and No preference.
Time Frame: Up to Study Week 24
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 Milligrams (mg) + RPV LA 900 mg (Q8W)
Number analyzed (Participants) | 51
Participants
  Injections in the buttock | 29
  Injections in the thigh | 17
  No preference | 5

34. Secondary Outcome: Number of Participants With Their Treatment Preference as Assessed Using Preference Questionnaire for CAB LA + RPV LA Q4W Arm
Description: A preference questionnaire was used to assess participant's preference for the thigh injections compared with the gluteal injections. The "Preference" questionnaire included a single item question evaluating preference of HIV treatment. Participants were required to provide their response to Question, which stated "Which injection site do you prefer". The responses included Injections in the buttock, Injections in the thigh, Other and No preference.
Time Frame: Up to Study Week 20
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 400 mg + RPV LA 600 mg (Q4W)
Number analyzed (Participants) | 61
Participants
  Injections in the buttock | 39
  Injections in the thigh | 17
  No preference | 5

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected up to 16 weeks during Thigh Injection Phase and from Week 16 to Week 24 during Return to Gluteal Injection Phase
Description: All-cause mortality, Non-SAEs and SAEs were reported for the sub-study Safety Population which included all randomized participants who received at least one CAB and/or RPV thigh injection. AEs were presented phase-wise.
Groups:
- CAB LA 600 mg + RPV LA 900 mg Q8W-Thigh Injection Phase: Participants received an IM injection of CAB LA 600 mg on one lateral thigh and RPV LA 900 mg into the opposite lateral thigh on Day 1 in every 8 weeks (Q8W) for a total of 16 weeks during Thigh Injection Phase.
- CAB LA 400 mg + RPV LA 600 mg (Q4W) -Thigh Injection Phase: Participants received an IM injection of CAB LA 400 mg on one lateral thigh and RPV LA 600 mg into the opposite lateral thigh on Day 1 in every 4 weeks (Q4W) for a total of 16 weeks Thigh Injection Phase
- CAB LA 600 mg + RPV LA 900 mg Q8W- Gluteal Injection Phase: Participants received first IM gluteal injection (at Week 16) of CAB LA 600 mg + RPV LA 900 mg during the return to Gluteal Injection Phase and subsequent gluteal injection occurred after Q8W.
- CAB LA 400 mg + RPV LA 600 mg (Q4W) - Gluteal Injection Phase: Participants received first IM gluteal injection (at Week 16) of CAB LA 400 mg + RPV LA 600 mg during the return to Gluteal Injection Phase and subsequent gluteal injection occurred after Q4W.
Arm/Group | CAB LA 600 mg + RPV LA 900 mg Q8W-Thigh Injection Phase | CAB LA 400 mg + RPV LA 600 mg (Q4W) -Thigh Injection Phase | CAB LA 600 mg + RPV LA 900 mg Q8W- Gluteal Injection Phase | CAB LA 400 mg + RPV LA 600 mg (Q4W) - Gluteal Injection Phase
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/64 | 0/51 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/64 | 1/51 | 0/61
Other Adverse Events (participants affected / at risk) | 38/54 | 46/64 | 6/51 | 11/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA 600 mg + RPV LA 900 mg Q8W-Thigh Injection Phase (N=54) | CAB LA 400 mg + RPV LA 600 mg (Q4W) -Thigh Injection Phase (N=64) | CAB LA 600 mg + RPV LA 900 mg Q8W- Gluteal Injection Phase (N=51) | CAB LA 400 mg + RPV LA 600 mg (Q4W) - Gluteal Injection Phase (N=61)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA 600 mg + RPV LA 900 mg Q8W-Thigh Injection Phase (N=54) | CAB LA 400 mg + RPV LA 600 mg (Q4W) -Thigh Injection Phase (N=64) | CAB LA 600 mg + RPV LA 900 mg Q8W- Gluteal Injection Phase (N=51) | CAB LA 400 mg + RPV LA 600 mg (Q4W) - Gluteal Injection Phase (N=61)
Injection site pain (General disorders) | 38 (110) | 43 (163) | 3 (4) | 9 (17)
Injection site discomfort (General disorders) | 3 (6) | 5 (8) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 5 (5) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT05896761/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT05896761/SAP_001.pdf